CLINICAL TRIAL: NCT06385093
Title: Efficacy and Safety of Eldecalcitol in Preventing Glucocorticoid-induced Bone Loss in Rheumatoid Arthritis Patients (ELEGANT)
Brief Title: A Study on the Prevention and Treatment of GIOP With Eldecalcitol
Acronym: ELEGANT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese SLE Treatment And Research Group (Other)
Collaborators: Beijing Life oasis public service center (Unknown)
Responsible Party: Principal Investigator, Mengtao Li, Professor and Director, Rheumatology and Immunology Department, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDR-IIS-003
Record Dates: First submitted 2024-04-09; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis; Osteoporosis; Osteopenia
Keywords: Rheumatoid Arthritis; Osteoporosis; Randomized Controlled Trial; Glucocorticoids; Eldecalcitol
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoporosis; Bone Diseases, Metabolic | interventions — eldecalcitol; alfacalcidol; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eldecalcitol (Experimental): Participants receive oral eldecalcitol 0.75μg daily for 12 months
  Interventions: Drug: Eldecalcitol capsules
- Alfacalcidol + calcium carbonate (Active Comparator): Participants receive oral calcitriol 0.5μg daily and 1.5g calcium carbonate daily for 12 months
  Interventions: Drug: Alfacalcidol tablets; Drug: Calcium carbonate tablets

INTERVENTIONS:
Drug: Eldecalcitol capsules — Oral eldecalcitol 0.75μg daily
  Other Names: Edirol
  Arms: Eldecalcitol
Drug: Alfacalcidol tablets — Oral Alfacalcidol 0.5μg daily
  Arms: Alfacalcidol + calcium carbonate
Drug: Calcium carbonate tablets — 1.5g Calcium carbonate daily
  Arms: Alfacalcidol + calcium carbonate

SUMMARY:
The study will be a multi-center, randomized, open label, parallel trial conducted in rheumatoid arthritis patients treated with glucocorticoids. After signing the informed consent, all patients will be screened as per the inclusion and exclusion criteria. Estimated 314 eligible patients will be enrolled. The enrolled patients will be randomly assigned to either Eldecalcitol group or Alfacalcidol group in a 1:1 ratio and followed up for 12 months. On-site follow up visits will be conducted at Month 6 and 12 after enrollment. The study is designed to evaluate the efficacy and safety of Eldecalcitol in preventing glucocorticoid-induced bone loss in rheumatoid arthritis patients.

DETAILED DESCRIPTION:
After having signed informed consent (Day 0), the patients will be screened for enrollment. About 314 eligible patients will be enrolled in this study. The background information of eligible patients including demographic characteristics, history of present illness, medical history, treatment history, etc., related questionnaire, baseline bone mineral density (BMD), X-ray examination result, High Resolution-Peripheral Quantitative Computed Tomography (HR-pQCT) examination result, quantitative ultrasound (QUS) examination result and lab test result will be collected at Day 0. After enrollment, the following information will be collected at 6 months and/or 12 months: related questionnaire, BMD, X-ray examination result, HR-pQCT examination result, QUS examination result and lab test result, medication adherence and AE information.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult rheumatoid arthritis patients(≥18 years) who fulfilled the 1987 American College of Rheumatology (ACR) criteria or the 2010 ACR/European League Against Rheumatism (EULAR) criteria.
* 2. Had been taking 5-10 mg oral prednisolone (or equivalent) daily glucocorticoids for longer than 3 months at screening and were expected to receive glucocorticoids for at least another 12 months.
* 3. Ambulant outpatients
* 4. Written informed consent

Exclusion Criteria:

* 1. BMD T<-3.0 measured by DXA at screening
* 2. Vertebral, hip, proximal humerus, pelvis, or distal forearm fragility fracture history
* 3. Any severe bone disorder or deformation at the lumbar spine that would affect DXA measurement
* 4. Primary hyperparathyroidism, Cushing's syndrome, hyperthyroidism, gonadal insufficiency, osteogenesis impotence, poorly controlled diabetes mellitus (HbA1c>9%), or other diseases that can affect bone metabolism
* 5. Had injected bisphosphonate once or more within 3 years before entering the study; or had received oral bisphosphonate for 6 months or more in the 3 years prior to study entry; or had received parathyroid hormone once or more in the 3 years before entering the study; or received 2 weeks or more of calcitonin or vitamin K or selective estrogen receptor modulator or hormone replacement therapy or traditional Chinese medicine for osteoporosis within 2 months prior to study entry; or received active vitamin D within 2 weeks prior to study entry; or received subcutaneous anti-RANKL antibody at any time prior to study entry
* 6. Urolithiasis at screening or had a history of urolithiasis
* 7. Hypercalcemia (serum calcium >10.4 mg/dL), or hypercalciuria (fasting morning urine calcium/creatinine >400 mg/gCr or 24h urine calcium >300mg), or had serum creatinine levels above the reference range
* 8. Severe liver disease such as cirrhosis or serious heart disease such as severe heart failure
* 9. Active malignant tumors or a history of malignant tumors within 5 years before informed consent obtained
* 10. History of allergy to vitamin D
* 11. Pregnant women or female patients planning to become pregnant during the study
* 12. Other inappropriate situations judged by investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline to month 12 in lumbar spine (L1-4) bone mineral density (BMD) | Baseline and 12 months
  BMD will be measured using dual energy x-ray absorptiometry (DXA). Images will be analyzed by blinded independent central review.

SECONDARY OUTCOMES:
Percent change from baseline to month 6 in lumbar spine (L1-4) BMD | Baseline and 6 months
  BMD will be measured using DXA. Images will be analyzed by blinded independent central review.
Percent change from baseline in total hip BMD | Baseline, 6 months and 12 months
  BMD will be measured using DXA. Images will be analyzed by blinded independent central review.
Percent change from baseline in femoral neck BMD | Baseline, 6 months and 12 months
  BMD will be measured using DXA. Images will be analyzed by blinded independent central review.
Percent change from baseline to month 12 in broadband ultrasound attenuation (BUA) and speed of sound (SOS) measured by quantitative ultrasound (QUS) | Baseline and 12 months
  Broadband ultrasound attenuation (BUA) and speed of sound (SOS) will be measured by quantitative ultrasound (QUS).
Percent change from baseline in Procollagen Type 1 N-telopeptide (P1NP) | Baseline, 6 months and 12 months
  Serum P1NP will be tested
Percent change from baseline in Type 1 Collagen C-telopeptide (CTX) | Baseline, 6 months and 12 months
  Serum CTX will be tested
Percentage of patients diagnosed with osteoporosis at month 12 | Baseline and 12 months
Incidence of new vertebral fracture | Baseline and 12 months
  New vertebral fracture will be confirmed by the lateral X-ray of thoracic/lumbar vertebrae
Change from baseline in Quality of Life assessed using EQ-5D-5L | Baseline, 6 months and 12 months
  The EQ-5D-5L represents a global quality of life measure that includes multiple components potentially impacted by the anti-anginal treatments being examined. The EQ-5D-5L score includes questions on mobility, self-care, usual activities, anxiety/depression, and pain/discomfort on a 5-point scale: 1=No Problem, 2=Slight Problem, 3=Moderate Problem, 4=Severe Problem, 5=Extreme Problem or Inability. 0, 1, and negative values corresponding to death, full health, and health states worse than death, respectively. Higher scores indicated greater levels of problems across each of the five dimensions.
Change from baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) | Baseline, 6 months and 12 months
  Physical function was assessed by HAQ-DI. It consisted of at least 2 questions per category, participant reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week rated on a 4-point scale where 0 = no difficulty; 1 = some difficulty; 2 = much difficulty; 3 = unable to do. Overall score was computed as the sum of category scores and divided by the number of categories answered, ranging from 0 to 3, where 0 = no disability and 3 = unable to do, high-dependency disability.
Change from baseline in Disease Activity Score for 28 Joints -C-Reactive Protein (DAS28--CRP) Score | Baseline, 6 months and 12 months
  DAS28 is a composite score that includes 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); General health (GH) assessment by the participant assessed from the ACR rheumatoid arthritis (RA) core set questionnaire (participant global assessment) in 100 mm visual analog scale (VAS). Marker of inflammation assessed by the high sensitivity C-reactive protein (hs-CRP) in mg/L. The DAS28 score provides a number indicating the current disease activity of the RA. DAS28 total score ranges from 2-10. A DAS28 score above 5.1 means high disease activity, whereas a DAS28 score below 3.2 indicates low disease activity and a DAS28 score below 2.6 means disease remission.
Percent change from baseline to month 12 in volumetric bone mineral density (vBMD) measured by High Resolution-Peripheral Quantitative Computed Tomography (HR-pQCT) | Baseline and 12 months
  The vBMD includes several individual parameters as total volumetric bone mineral density (Tt.vBMD), trabecular volumetric bone density (Tb.vBMD), and cortical volumetric density (Ct.vBMD) which all in milligram/cubic centimetre.
Percent change from baseline to month 12 in bone microarchitecture measured by High Resolution-Peripheral Quantitative Computed Tomography (HR-pQCT) | Baseline and 12 months
  The bone microarchitecture include several individual parameters as trabecular bone volume fraction (BV/TV) in %, trabecular number (Tb.N) in 1/millimeter, trabecular thickness (Tb.Th) in millimeter, trabecular separation (Tb.Sp) in millimeter, cortical thickness(Ct.Th) in millimeter, and cortical porosity (Ct.Po) in %.
Percent change from baseline to month 12 in bone geometry measured by High Resolution-Peripheral Quantitative Computed Tomography (HR-pQCT) | Baseline and 12 months
  The bone geometry include several individual parameters as total bone cross-sectional area (Tt.Ar), cortical area (Ct.Ar), and trabecular area (Tb.Ar) which all in square millimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Mengtao Li, MD, Principal Investigator — Peking Union Medical College Hospital; Weibo Xia, MD, Principal Investigator — Peking Union Medical College Hospital; Ying Jiang, MD, Study Director — Peking Union Medical College Hospital
Locations (7):
- China (7):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Aerospace Central Hospital, Beijing, Beijing Municipality
  - Beijing Luhe hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Shijingshan Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Beijing Shunyi hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality